CLINICAL TRIAL: NCT07116980
Title: Biological and Psychological Markers After Trancranial Electrical Stimulation in Adults With Generalized Anxiety Disorder
Brief Title: Biological and Psychological Markers After Intervention in Adults With GAD
Acronym: AnsitDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69019123.3.0000.5327
Record Dates: First submitted 2025-06-18; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Anxiety
Keywords: anxiety; tDCS; IL-6; Cortisol; HRV; EEG
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel-group, simulation-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher will receive equipment already programmed by a research assistant, therefore, the researcher who will deliver the tDCS to perform the stimulation will not know the programmed stimulation. Patients will be instructed to discuss aspects of treatment with the respective investigator. Two independent assessors who will not participate in consultations where guidance on the use of tDCS will be provided will be trained to assess follow-up outcomes. Patients will not know the type of intervention received, as the sham condition produces a stimulus, but without the expected effects. Blinding will be evaluated at the end of treatment using a standardized instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- responds to the placebo effect Intervention: Transcranial Direct Current Stimulation - tDCS (Placebo Comparator): Patients will receive tDCS stimulation treatment dorsolateral prefrontal cortex. According to the 10-20 EEG system, the anode will be placed on the left F3 and the cathode on the contralateral F4.
  Placebo stimulation uses a current of 2 milliamps for the first 30 seconds and again for the last 30 seconds. The tDCS application time will be 20 minutes Device: s-tDCS - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it
  Device: a-tDCS
  - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it
  Interventions: Device: 'Transcranial Direct Current Stimulation - tDCS
- No placebo effect responds Intervention: Transcranial Direct Current Stimulation - tDCS (Active Comparator): Patients will receive tDCS stimulation treatment dorsolateral prefrontal cortex According to the 10-20 EEG system, the anode will be placed on the left F3 and the cathode on the contralateral F4.
  Active stimulation uses a current of 2 milliamps for 20 minutes. Device: s-tDCS - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it
  Device: a-tDCS
  - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it
  Interventions: Device: 'Transcranial Direct Current Stimulation - tDCS

INTERVENTIONS:
Device: 'Transcranial Direct Current Stimulation - tDCS — Participants will receive by trained personnel, transcranial direct current stimulation (tDCS) targeting the dorsolateral prefrontal cortex (DLPFC). According to the international 10-20 EEG system, the anodal electrode will be placed over the left F3 position and the cathodal electrode over the right F4 position. Active stimulation will be delivered using a constant current of 2 milliamperes (mA) for 20 minutes per session. The intervention will consist of twelve consecutive daily sessions (Monday to Friday), totaling four week of treatment. A certified tDCS device will be used, programmed to deliver a ramp-up and ramp-down period of 30 seconds.
  In the sham condition, the same electrode montage will be used; however, the device will automatically ramp down the current after 30 seconds, mimicking the initial tingling sensation without producing lasting neuromodulatory effects. This sham protocol is commonly used to ensure participant blinding in tDCS studies.

SUMMARY:
This clinical trial inestigates the effects of transcranial direct current stimulation (tDCS) on anxiety symptoms in adult women with clinically relevant anxiety levels. The intervention involves the application of low-intensity electrical current over the left dorsolateral prefrontal cortex (DLPFC) across twenty consecutive sessions. Participants are randomly assigned to either an active or sham stimulation group in a double-blind design. The study aims to evaluate changes in anxiety symptoms, emotional regulation, and physiological and molecular markers, including EEG activity, heart rate variability (HRV), and salivary levels of cortisol and interleukin-6 (IL-6) plasma. The findings are expected to support the development of complementary, low-cost, and non-pharmacological strategies for anxiety management.

DETAILED DESCRIPTION:
Anxiety is one of the biggest causes of disability in the world, and many patients do not respond to conventional treatments. Due to this situation, studies were carried out to understand better understand the mechanisms of psychiatric disorders, and one of the alternatives found was the non-invasive brain stimulation with transcranial direct current (tDCS). The project in question aims to evaluate the effectiveness of tDCS-based intervention in adults with anxiety, comparing with a control group. The results will be measured through questionnaires and tests cognitive effects, as well as analyzes of physiological data and inflammatory markers. The study will be done through an experimental and a control group, with 49 men and women in each group. All data will be collected at the Neuromodulation laboratory at Hospital de Clínicas de Porto Alegre, under the coordination of Professor Wolnei Caumo. Participants will be recruited through previously registered patients on Neuromodulation laboratory at Hospital de Clínicas de Porto Alegre database, and the inclusion criteria and exclusion will be defined according to values of anxiety scales and other characteristics of health. The entire process will be conducted safely. Participants in the experimental and control will have their data collected on the first and last day of the intervention. Each participant will receive a placebo or control intervention of 20 sessions, between the first and the last, and will be blinded between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults under the age of 18;
* GAD-7 ≥ 10
* Possibility of being present on previously agreed days.

Exclusion Criteria:

* Being in psychopharmacological treatment for depression;
* HAM-D≥23 scale;
* have a self-reported severe disorder (psychosis, schizophrenia, substance abuse, major depression);
* having had seizures and epilepsy;
* having presented substance use disorder (except Tobacco) in the last 6 months or Suicidal Ideation in the last 6 months;
* being pregnant or breastfeeding;
* have suffered any type of brain injury or surgery, heart disease or cranial defect.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Symptoms as Assessed by the GAD-7 Scale | 1 month
  Change in anxiety symptoms will be assessed by the total change in the GAD-7 score, a 7-item self-administered scale that measures the severity of anxiety symptoms. Scores range from 0 to 21, with higher scores indicating greater anxiety severity.

SECONDARY OUTCOMES:
Change in the Anxiety Sensitivity Index-Revised (ASI-R) Total Score | 1 month
  The change in anxiety sensitivity will be assessed by the total change in the Anxiety Sensitivity Index-Revised (ASI-R) score, a 36-item questionnaire that measures the fear of anxiety-related sensations. Higher scores indicate greater anxiety sensitivity.
Change in Pain Intensity as Measured by the Central Sensitization Inventory (CSI) score | 1 month
  The change in pain intensity will be assessed by the Central Sensitization Inventory (CSI), a 25-item self-report questionnaire that assesses common symptoms associated with central sensitization. The scale is scored from 0 to 100, with higher scores indicating higher levels of central sensitization.
Change in Subjective Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI) score | 1 month
  The change in subjective sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI) score. The PSQI is a self-rated questionnaire that assesses sleep quality over the last month. The scale includes seven component scores, and a global score is derived, ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Change in Absolute Alpha Band Power (8-12 Hz) at Electrode Site [F3/F4/C3/C4/P3/P4] as Assessed by Electroencephalogram (EEG). | 1 month
  Absolute alpha band power will be calculated from resting EEG recordings and expressed in µV²/Hz. Recordings will be acquired from the [specific electrode site] electrode.
Change in Heart Rate Variability (HRV) as Assessed by the Standard Deviation of NN Intervals (SDNN) | 1 month
  SDNN will be collected from 3-minute resting recordings and expressed in milliseconds (ms).
  This specifies the exact HRV metric (SDNN) and its unit, making it clear and quantifiable
Change in Interhemispheric Absolute Alpha Band Power Asymmetry (8-12 Hz) Between [F3 and F4 / C3 and C4 / P3 and P4] as Assessed by Electroencephalogram (EEG) | 1 month
  Interhemispheric absolute alpha band power asymmetry will be calculated from resting EEG recordings and expressed as a ratio. Recordings will be acquired from [F3 and F4 / C3 and C4 / P3 and P4] electrode pairs.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
Given the potential for this study to be extended in future research protocols involving different variables, the current stage is not appropriate for public data sharing.

REFERENCES:
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Chalmers JA, Quintana DS, Abbott MJ, Kemp AH. Anxiety Disorders are Associated with Reduced Heart Rate Variability: A Meta-Analysis. Front Psychiatry. 2014 Jul 11;5:80. doi: 10.3389/fpsyt.2014.00080. eCollection 2014. PMID 25071612
- [Background] Dedoncker J, Brunoni AR, Baeken C, Vanderhasselt MA. A Systematic Review and Meta-Analysis of the Effects of Transcranial Direct Current Stimulation (tDCS) Over the Dorsolateral Prefrontal Cortex in Healthy and Neuropsychiatric Samples: Influence of Stimulation Parameters. Brain Stimul. 2016 Jul-Aug;9(4):501-17. doi: 10.1016/j.brs.2016.04.006. Epub 2016 Apr 12. PMID 27160468
- [Background] Palm U, Hasan A, Strube W, Padberg F. tDCS for the treatment of depression: a comprehensive review. Eur Arch Psychiatry Clin Neurosci. 2016 Dec;266(8):681-694. doi: 10.1007/s00406-016-0674-9. Epub 2016 Feb 3. PMID 26842422
- [Background] Shiozawa P, Leiva AP, Castro CD, da Silva ME, Cordeiro Q, Fregni F, Brunoni AR. Transcranial direct current stimulation for generalized anxiety disorder: a case study. Biol Psychiatry. 2014 Jun 1;75(11):e17-8. doi: 10.1016/j.biopsych.2013.07.014. Epub 2013 Aug 16. No abstract available. PMID 23958182
- [Background] Brunoni AR, Vanderhasselt MA. Working memory improvement with non-invasive brain stimulation of the dorsolateral prefrontal cortex: a systematic review and meta-analysis. Brain Cogn. 2014 Apr;86:1-9. doi: 10.1016/j.bandc.2014.01.008. Epub 2014 Feb 8. PMID 24514153